CLINICAL TRIAL: NCT05294952
Title: Levels of Co-inhibitory Receptors (TIM-3,LAG-3 and TIGIT)in Preeclampsia Patients
Brief Title: co Ihibtory Receptor in Preeclampsia
Acronym: asd
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Ibrahim Sayed, real time PCR, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: zisdas
Record Dates: First submitted 2022-03-04; First posted 2022-03-24 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Pre-Eclampsia
Keywords: coinhibtory receptor
MeSH Terms: conditions — Pre-Eclampsia | interventions — Real-Time Polymerase Chain Reaction; Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Intervention Model Description: preeclasmpsia pregnant women and normal pregnant women
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preeclampsiapregnant women (Experimental): Inclusion criteria
  A total of 41 women in third trimester pregnancy complicated with PE showing:
  * Blood pressure ≥140/90 mmHg and
  * Proteinuria ≥300 mg/24 hours with or without
  * Edema in pregnant woman after week 20 of gestation (American Congress of Obstetricians and Gynecologists (ACOG2013) (17)
  B-Exclusion criteria
  * Patients with autoimmune, acute inflammatory, and chronic diseases, are excluded from the study.
  Interventions: Genetic: real time PCR
- normal pregnant women (No Intervention): This will include age matched 41 normal pregnant women in their third trimester of pregnancy with normal blood pressure, absence of proteinuria, and without any other systemic or endocrine disorder.

INTERVENTIONS:
Genetic: real time PCR — diagnostic test
  Other Names: ELISA
  Arms: preeclampsiapregnant women

SUMMARY:
Preeclampsia is a form of hypertensive pregnancy disorder with multiorgan involvement. It is characterized by new-onset hypertension and proteinuria after 20 weeks' gestation in a woman whose blood pressure was normal before pregnancy. The condition may be serious and is a leading cause of preterm birth (before 37 weeks of pregnancy). If it is severe enough it may affect the brain function, causing seizures or coma, this is called eclampsia

DETAILED DESCRIPTION:
T lymphocytes, as well as their regulatory subpopulations could possibly possess a part in PE . The changes in T cell subsets that may be seen in preeclampsia include low Treg activity, a shift toward Th1 responses, and the presence Th17 lymphocytes. B cells can participate in the pathophysiology of preeclampsia by producing autoantibodies against adrenoreceptors and autoantibodies that bind the AT1-R (angiotensin II type I receptor)

TH17 cells are a distinctive lineage of TCD4+ cells, which are distinguished by producing a number of effective molecules such as IL-17, which is the most important cytokine produced by these cells . IL-17 is capable of inducing the production of several cytokines, such as tumor necrosis factor alpha (TNF-α) and IL-1β which possess significant parts in PE pathophysiology .

Regulatory T lymphocytes CD4+ CD25bright are known to play an important role in the development and maintenance of tolerance in peripheral tissues . They express high level of CD25 (IL-2Ra) as well as cytotoxic T-lymphocyte antigen 4 (CTLA4) and the transcription factor Foxp3 .

It was proposed that regulatory T cells (Tregs) are responsible for mediating maternal tolerance for the fetus and their counts were found to be higher in normal pregnancies However, the role of T reg cells in the development of preeclampsia remains controversial, being decreased in some studies .) and of comparable frequencies to normal pregnancy in others (Hu et, 2008). Tregs suppress maternal immune cells through the secretion of inhibitory cytokines, such as interleukin (IL)-10 and transforming growth factor beta (TGF-β) .

systemic endothelial dysfunction, such as disturbed coagulation function, could be intensified through immune activation, resulting in inflammation and the disturbance of regulatory T (Treg) and Th17 cell balance, and contributing to further activation of the maternal immune responses .

Co-inhibitory-receptors such as CTLA-4 (cytotoxic T-lymphocyte-associated protein , LAG-3 (lymphocyte activation gene 3; or CD223), TIM-3 (T-cell immunoglobulin and mucin domain-containing 3), PD-1 (PDCD1; programmed cell death 1), and TIGIT (T-cell immunoreceptor with Ig and ITIM domains) are key factors in maintaining immune homeostasis and play a central role in regulating autoimmune diseases .

These receptors regulate T-cell responses by inhibiting effector T-cell activation directly by promoting the suppressive function of regulatory T-cells (Tregs) and affecting antigen presentation. These cell surface molecules are expressed on activated immune cells (T-cells, B cells, natural killer [NK] cells, some myeloid cells) that regulate the inflammatory and autoimmune responses through a negative feedback mechanism. Malfunction of their crucial role or decreased receptor levels can lead to excessive immune activation and autoimmunity .

While augmented effector T-cell activation plays a major role in preeclampsia pathogenesis, insufficient co-inhibitory signals might promote preeclampsia development and progression. Some studies have also shown that multiple co-inhibitory-molecules, e.g., TIM-3, LAG-3, and TIGIT, predominantly regulate the effector T-cell responses within the tissue where their responses are executed . Based on the previous findings on the important role of the co-inhibitory molecules in regulating autoimmunity and cancer immunity, it might be assumed that they also play a role in preeclampsia development and/or progression.

ELIGIBILITY:
Inclusion Criteria:

* total of 41 women in third trimester pregnancy complicated with PE showing:

  * Blood pressure ≥140/90 mmHg and
  * Proteinuria ≥300 mg/24 hours with or without
  * Edema in pregnant woman after week 20 of gestation (American Congress of Obstetricians and Gynecologists (ACOG2013) (17)

Exclusion Criteria:

* B-Exclusion criteria • Patients with autoimmune, acute inflammatory, and chronic diseases, are excluded from the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female
Enrollment: 82 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-02-03 (Estimated); Study Completion 2025-11-04 (Estimated)

PRIMARY OUTCOMES:
early detection of preeclampsia | 1year
  detection levels of co inhibtory receptor

IPD SHARING:
Plan to Share IPD: No